CLINICAL TRIAL: NCT03823599
Title: A Pilot Study on the Feasibility of Alcohol Brief Intervention Plus Personalized Mobile Chat-based Intervention to Reduce Alcohol Misuse in an Emergency Department in Hong Kong
Brief Title: Alcohol Brief Intervention Plus Personalized Mobile Chat-based Intervention to Reduce Alcohol Misuse in an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pilot alcohol study (AED)
Record Dates: First submitted 2019-01-27; First posted 2019-01-30 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Use Disorder
Keywords: chat-based intervention; alcohol brief intervention; Alcohol misuse; Accident & Emergency Department; AUDIT; instant messaging
MeSH Terms: conditions — Alcoholism; Emergencies | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Alcohol brief intervention+mobile chat-based instant messages
  Interventions: Behavioral: Mobile chat-based instant messages; Behavioral: Alcohol brief intervention
- control group (Active Comparator): Alcohol brief intervention
  Interventions: Behavioral: Alcohol brief intervention

INTERVENTIONS:
Behavioral: Mobile chat-based instant messages — Subjects in the active arm study will receive 5-minute face-to-face ABI, alcohol leaflet from Department of Health (DH) plus continuous interactive chat-based intervention for 1 month as an extension of alcohol brief intervention at baseline
  Arms: Intervention group
Behavioral: Alcohol brief intervention — The Control group will receive face-to-face ABI plus an alcohol leaflet from DH.

SUMMARY:
This project focuses on patients in AED. Objectives of this project are:

1. To examine the factors associated with alcohol drinking and alcohol use disorder
2. To examine the effect of face-to-face alcohol brief intervention on drinking reduction
3. To examine the effect of a continuous interactive chat-based intervention via "WhatsApp" on drinking reduction
4. To explore the perception of face-to-face alcohol brief intervention
5. To explore the perception of continuous interactive chat-based intervention via instant messaging mobile application "WhatsApp"

DETAILED DESCRIPTION:
According to the Department of Health, a local epidemiological study was conducted in 2001 and showed that about one in ten of all motor vehicle deaths were associated with alcohol consumption. Also, the statistics from the Transportation department showed that 874 vehicle accidents resulting in personal injury were related to alcohol misuse, which included 24 fatal cases between the period of 2000 and 2010. With the aforementioned statistics supported, the hospital Accident and Emergency Department (AED) serves as the most important entrance and safeguard to the healthcare system for the public, since victims of traffic accidents or violence related to heavy drinking are frequently encountered in AED, this serves as an ideal place for provision of initial alcohol intervention and further stabilization related to alcohol problem of patients. Although AED is a hectic environment with very high patients turnover, substantial evidence had shown feasibility and efficacy of Alcohol Brief Intervention (ABI) in reducing patients' subsequent alcohol drinking. In oversea, multiple research had been done to show ABI were effective and feasible for reducing alcohol misuse, but the effect was not long lasting and lead to subsequent relapse. In addition to this, no further trial has been done to investigate the feasibility of implementing an RCT on evaluating the effect of ABI and continuous chat-based intervention on reducing alcohol consumption among patients in AED in Hong Kong.

According to the WHO, the standard ABI approach includes: giving feedback and information about the screening result and hazard of drinking; emphasizing the benefits of quit drinking and informing about alcohol problems; setting goal on reducing alcohol consumption; reviewing advice and ; giving encouragement. In this pilot study, a brief alcohol counselling using face-to-face ABI will be delivered together with continuous interactive chat-based intervention via instant messaging mobile application "WhatsApp" to those patients with AUDIT score ≥ 8, who are considered to have hazardous and harmful drinking problems according to the guideline.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong resident aged 18 to 65
2. scored ≥ 8 in the Alcohol Use Disorder Identification Test (AUDIT) in the past 12 months
3. able to communicate in Cantonese (including reading Chinese)
4. using a phone with instant messaging mobile application "WhatsApp" installed for communication.

Exclusion Criteria:

1. patients with communication barrier (either physically or cognitively)
2. currently participating in other alcohol treatment services or clinics
3. will be hospitalized immediate after A&E consultation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
change in unit of alcohol consumption in gram | at 3-month after baseline.
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 3-month after baseline.

SECONDARY OUTCOMES:
change in unit of alcohol consumption in gram | at 1-month after phase I
  Assessed by unit in gram and compare the alcohol consumption between intervention and control group at 1-month after phase I
change in episode of binge drinking measured by asking "Never", "less than a month", "two to four times a month", " two to three times a week" and "almost everyday" | at 1 and 3 months after phase I
  Defined by 5 [male] or 4 [female] in a row for binge drinking and compare the episode of binge drinking between intervention group and control at baseline, 1 and 3-month follow-up questionnaires
change in frequency of drinking by asking "Never", "less than a month", "two to four times a month", " two to three times a week" and "almost everyday" | at 1 and 3 months after phase I
  Compare the frequency of drinking between intervention group and control at baseline, 1 and 3-month follow-up questionnaires
attempt to reduce drinking measured by asking whether they have tried to reduce drinking at past month (yes or no) | at 1 and 3 months after phase I
  Compare the attempt to reduce drinking between intervention group and control group at baseline, 1 and 3-month follow-up questionnaires
change in confidence to reduce drinking measured by Likert scale (1-10) | at 1 and 3 months after phase I
  Score ranges from 0 to 10 with higher score indicates a high level. The score will be compared between intervention group and control group at baseline, 1 and 3-month follow-up questionnaires
Alcohol Problems Scale at 1 and 3-month follow-up | at 1 and 3 months after phase I
  The 14-item measure of alcohol-related personal, social, sexual, and legal problems (eg, being physically aggressive toward someone while under the influence of alcohol).The score will be compared between intervention group and control group at baseline, 1 and 3-month follow-up questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided